CLINICAL TRIAL: NCT03712514
Title: Dynamic Stabilization of the Upper Cervical Spine in a Cohort of Rugby's Players Via Ergometer (Cervistab©)
Brief Title: Behavior of the Upper Cervical Spine in Rugby Players
Acronym: Cervistab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the inclusion period ended on 23/09/2021
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9536; 2015-A00505-44 (Other: ANSM)
Record Dates: First submitted 2018-04-27; First posted 2018-10-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2021-12

CONDITIONS: Cervical Spine Destabilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rugby players (Other): Destabilization of the upper cervical spine with Cervistab
  Interventions: Other: Destabilization of the upper cervical spine by Cervistab
- Healthy non rugby players (Other): Destabilization of the upper cervical spine with Cervistab
  Interventions: Other: Destabilization of the upper cervical spine by Cervistab

INTERVENTIONS:
Other: Destabilization of the upper cervical spine by Cervistab — Simulate a situation of destabilization of the cervical spine with Cervistab

SUMMARY:
Rugby players are often exposed to destabilisation of the upper cervical spine.This kind of trauma may lead to dramatic injuries, due to lesion of spinal cord.

CerviStab© is a device which evaluate the bio-mechanical and neuromuscular behavior of the upper cervical spine in rugby situation.

The aim of this study, is to evaluate the dynamic stabilization of the upper cervical spine in reaction to unexpected impact.

ELIGIBILITY:
Inclusion Criteria:

* Rugby players at least since 5 years
* Amateurs or professionals players
* Able to play in rugby competition

Exclusion Criteria:

* Medical history of cervical spine injury requiring surgical intervention
* Active cervical symptomatology
* Medical history of migraine or epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Reproducibility of head movement amplitude measurements on healthy volunteers | Week 1
  Measurement in millimetres by "Cervistab" ergometer
Reproducibility of the measurement of mechanical resistance strength intensity produced by upper cervical spine muscles responding to destabilization on healthy volunteers | Week 1
  Measurement in decanewtons by "Cervistab" ergometer
Reproducibility of time until appearance of mechanical resistance strength produced by upper cervical spine muscles responding to destabilization on healthy volunteers | Week 1
  Measurement in milliseconds by "Cervistab" ergometer
Reproducibility of the time of response of upper cervical spine extensor muscles responding to destabilization on healthy volunteers | Week 1
  Measurement in milliseconds by "Cervistab" ergometer
Reproducibility of the amplitude of the response of upper cervical spine extensor muscles responding to destabilization on healthy volunteers | Week 1
  Measurement in decanewtons by "Cervistab" ergometer

SECONDARY OUTCOMES:
Comparison of biomechanical behaviour of upper cervical spine dynamic stabilization capacities between healthy volunteers and rugby players | Week 1
  Measurement by "Cervistab" ergometer
Comparison of neuromuscular behaviour of upper cervical spine dynamic stabilization capacities between healthy volunteers and rugby players | Week 1
  Measurement by "Cervistab" ergometer
Comparison of biomechanical behaviour of upper cervical spine dynamic stabilization capacities between resting and acute fatigue situations in rugby players subjects | Week 1
  Measurement by "Cervistab" ergometer
Comparison of neuromuscular behaviour of upper cervical spine dynamic stabilization capacities between resting and acute fatigue situations in rugby players subjects | Week 1
  Measurement by "Cervistab" ergometer
Comparison of biomechanical behaviour of upper cervical spine dynamic stabilization capacities between male rugby players and female rugby players | Week 1
  Measurement by "Cervistab" ergometer
Comparison of neuromuscular behaviour of upper cervical spine dynamic stabilization capacities between male rugby players and female rugby players | Week 1
  Measurement by "Cervistab" ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier university Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No